CLINICAL TRIAL: NCT01830647
Title: Non-interventional Local Study to Describe the Safety, Tolerability and Efficacy of Bevacizumab in Combination With Standard Chemotherapy Regimens as First Line in Patients With Metastatic Cancer of the Colon or the Rectum
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Cancer of the Colon or Rectum
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28411
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the safety and efficacy of first-line Avastin (bevacizumab) in combination with standard chemotherapy in routine clinical practice in patients with metastatic cancer of the colon and/or rectum. Patients will be followed for the duration of their treatment and a 30-day follow-up after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed carcinoma of the colon and/or rectum with evidence of metastases
* At least one measurable metastatic lesion (as per RECIST criteria)
* Life expectancy of > 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Clinically significant cardiovascular disease
* Ongoing treatment with aspirin (325 mg/day) or other medications known to predispose for gastrointestinal ulceration
* Participation in an investigational trial in the previous 3 months
* Pregnant or lactating women
* History of thrombotic or haemorrhagic disorders
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled hypertension
* Known hypersensitivity to Avastin and any of its excipients, or any of the chemotherapies
* Evidence of any disease or disorder that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer of the colon and/or rectum
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3.5 years

SECONDARY OUTCOMES:
Efficacy: Time to disease progression | approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Podgorica, Montenegro